CLINICAL TRIAL: NCT03301454
Title: Phase II Randomized Study Measuring the Interest of Pursuing or Not the CT for Non-progressive Patients With Metastatic Esophageal Squamous-cell Cancer After 6 Weeks of LV5FU2-paclitaxel Given After a 1st Line Fluoropyrimidine/Pt Salt CT
Brief Title: Study of the Interest of Pursuing or Not the Chemotherapy for Patients With Metastatic Esophageal Cancer
Acronym: E-DIS2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-DIS2-1705; 2017-003660-13 (EudraCT Number); 170757A-12 (Other: ANSM)
Record Dates: First submitted 2017-09-12; First posted 2017-10-04 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Esophageal Cancer, Squamous Cell
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Pursuit of chemotherapy.
  Interventions: Drug: pursuit of chemotherapy
- Arm B (No Intervention): Interruption of chemotherapy, best supportive care

INTERVENTIONS:
Drug: pursuit of chemotherapy — Treatment with LV5FU2 (5-FU, Calcium Levofolinate) - paclitaxel, regular tumor evaluation, best supportive care Other authorized treatment : usual paclitaxel pre-treatment consisting of Dexamethasone, Chlorpheniramine and ranitidine, at 15 and 1 day before the actual paclitaxel treatment
  Other Names: LV5FU2-paclitaxel CT
  Arms: Arm A

SUMMARY:
Phase II study, randomized, open-label, multicentric, willing to establish the benefit of pursuing chemotherapy beyond 6 weeks for non progressive patients. The study will proceed in two successive phases :

* non randomized phase in which all patients will undergo chemotherapy
* second phase in which only non progressive patients are going to be randomized ("discontinuation design"). Patients that will show progression in their disease during the first 6 weeks will be released of the study

DETAILED DESCRIPTION:
Initial phase: this part of the trial consist of 3 cycles of LV5FU2 (Bolus 5-FU 400mg/m² - 5-FU continuously during 46h: 3000 mg/m², calcium levofolinate 200 mg/m²) - paclitaxel (100 mg/m² at day 1) every 14 days. After 6 weeks,the phase will end with a check-up (clinical exam, tumor evaluation and biological test). Then, if the disease is non-progressive, the patient will proceed to the randomized phase.

Randomized phase:

* Arm A : pursuit of chemotherapy and best supportive care
* Arm B : interruption of chemotherapy and best supportive care

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from squamous-cell type esophageal cancer histologically proved
* Metastatic disease measurable according to RECIST criteria. Patients with metachronous metastasis and who have been treated with surgery (+/- radio chemotherapy concurrent or adjuvant chemotherapy) or exclusive radio chemotherapy, are eligible
* Patients who show progress under chemotherapy that associates a fluoropyrimidine with a platinum salt
* Man or woman over 18 years old
* ECOG performance status ≤ 2
* Adequate haematological, renal and hepatic functions : PNN ≥ 1500/ mm3; platelets ≥ 100 000/ mm3; Haemoglobin ≥ 9.0 g/dL; ALT and AST ≤ 2.5 ULN (≤ 5.0 in case of liver metastases); Total bilirubin ≤ 1.5 X ULN; Serum creatinine ≤ 1.5 ULN
* Efficient contraceptive method for both gender (if applicable), during the whole treatment period and the 6 months following the last treatment administration
* Affiliation to the National Social Security System
* With informed and signed consent

Inclusion Criteria for randomization:

* ECOG performance status ≤ 2
* Able to pursuit the LV5FU2-paclitaxel chemotherapy
* Non-progressive disease after the initial phase (first tumor exam at week 6)

Exclusion Criteria:

* Patients who received more than one line of chemotherapy for a metastatic disease
* Presence of other evolutive tumors
* Cerebral metastasis or other known brain tumors
* Severe liver failure
* Pernicious anemia or other anemia due to vitamin B12 defficiency
* Hypersensibility to an active substance or any other excipients of experimental drugs
* Every unstable chronicle diseases that can affect patient confidence or security
* Clinically significant active cardiac disease or myocardial infarction in the 6 previous months
* Patients with a known dihydropyrimidine dehydrogenase (DPD) deficiency
* Concomitant treatment with : sorivudin or analogs; prophylactic phenytoin
* Live attenuated vaccine within the 3 previous months
* Pregnant or breastfeeding women
* Unable to comply with the medical monitoring for geographic, social or mental issues
* Patient Under guardianship or tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Estimate the overall survival for patients suffering from Esophageal cancer | From date of randomization until the date of death from any cause, up to 8 months after the beginning of the treatment
  Non-progressive disease at and after 6 weeks of treatment until progression

SECONDARY OUTCOMES:
Estimate efficiency in term of overall survival, of pursuing chemotherapy | From date of randomization until the date of death from any cause, up to 8 months after the beginning of the treatment
  beyond 6 weeks of treatment compared to a group that interrupted the treatment at 6 weeks
Estimate the efficiency in term of progression-free of pursuing chemotherapy | From date of randomization until the date of first documented progression or date of death from any cause, up to 8 months after the beginning of the treatment
  beyond 6 weeks of treatment
Estimate the rate of non progressive patients | From date of inclusion until the date of the end the 6 firsts weeks of treatment
  after the 6 firsts weeks of treatment
Estimate the overall survival of the whole study population | From date of inclusion until the date of death from any cause, up to 8 months after the beginning of the treatment
  beyond the inclusion
Measure the toxicity of chemotherapy | from baseline up to 12 months
  during the initial treatment phase compared to the 2 treatment arms after randomization
Estimate the consequences of pursuing chemotherapy | From date of randomization until the date of first documented progression or date of death from any cause, up to 8 months after the beginning of the treatment
  beyond 6 weeks of treatment in term of time until degradation of life quality and in term of overall benefits

CONTACTS AND LOCATIONS:
Overall Officials: Farid EL HAJBI, MD, Principal Investigator — Centre Oscar Lambret
Locations (7):
- France (7):
  - Centre Hospitalier Universitaire, Amiens
  - Centre Paul Papin, Angers
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre René Gauducheau, Nantes
  - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, Plérin
  - Centre Eugène Marquis, Rennes

IPD SHARING:
Plan to Share IPD: No